CLINICAL TRIAL: NCT05607147
Title: Rutgers Pilot for Pragmatic Return to Effective Dental Infection Control Through Triage and Testing (PREDICT)- Dental Health Care Workers
Brief Title: Rutgers Pilot for Dental Health Care Worker SARS-CoV-2 Testing
Acronym: PREDICT-DHCW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2020002896; X01DE030407 (Other: NIDCR)
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: SARS-CoV2 Infection
Keywords: Dental Healthcare Worker; Testing; Seroprevalence; Perception of Safety; Adoption of risk mitigation practice
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Pilot study to assess feasibility of testing dental healthcare workers for seropositivity and antigen positivity for SARS-CoV-2 (Rapid Antigen point-of-care testing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SARS-CoV-2 testing (Other): There is only one arm in this study- the study is a non-randomized pilot. All the subjects will be tested for SARS CoV 2 viral Antigen and antibody to the virus as described.
  Interventions: Device: Testing for SARS CoV2 Antigen and Antibody

INTERVENTIONS:
Device: Testing for SARS CoV2 Antigen and Antibody — Antigen testing: Rapid Antigen testing (Point-of-care) Antibody testing: ELISA testing of microsampling 'finger-prick' specimen DHCW Survey for adoption of risk mitigation practices and for perceptions of safety

SUMMARY:
10 asymptomatic DHCWs in the Oral Medicine clinic, Rutgers School of Dental Medicine, with no history of documented COVID-19 infection or viral exposure, were enrolled in a study that interrogated DHCWs' perceptions of safety and adoption of risk mitigation behavior. Following a baseline survey, finger-prick blood samples were collected twice two weeks apart using an innovative microsampling technique that replaces the need for venipuncture. Samples were processed using an in-house ELISA assay to detect IgM and IgG directed against the Receptor Binding Domain (RBD) of the Spike protein. Weekly Rapid Antigen testing of nasal swab specimens was used to document Antigen negativity during the study.

DETAILED DESCRIPTION:
10 asymptomatic DHCWs in the Oral Medicine clinic, Rutgers School of Dental Medicine, with no history of documented COVID-19 infection or viral exposure, were enrolled in the DHCW arm of the study. The DCHWs underwent triage that included self-reported symptoms, temperature check and obtaining a pulse oximeter reading at every study time-point (See DHCW Arm in Results Section). Weekly Rapid Antigen testing of nasal swab specimens was used to document Antigen negativity during the study (BD Veritor Plus Analyzer, BD Sciences). The DHCWs' perceptions of safety and adoption of risk mitigation behavior were interrogated. Following a baseline survey, finger-prick blood samples were collected twice two weeks apart using avolumentric absorptive microsampling with a Neoteryx Mitra cartridge device (https://www.neoteryx.com) device that allows for self-sampling by non-specialized personnel (https://doi.org/10.1101/2021.07.09.21260266). Briefly, this microsampler allows for volumentric absorption of 10-30 μl of blood depending on selected size. Following the collection, microsamplers were dried and kept within the protective cassettes at room temperature for maximum period of 2 weeks from the collection date. Each microsampler tip (20µl in the present study) was added to 200 μl VAMS extraction buffer (1x PBS (Corning) supplemented with 1% bovine serum albumin (Roche Diagnostics, Mannheim, Germany) and 0.5% Tween20 (Sigma, MO, USA) in a 1 ml deep-well 96 well plate (Greiner bio-one-780261). The plate was then covered with an adhesive seal and incubated 16 hours at 40C on a shaker at 250 rpm. The resulting eluates were heat inactivated at 560C for 60 minutes and centrifugation to collect the supernatant (eluate). Eluates were further processed for an in-house ELISA assay to detect IgM and IgG directed against the Receptor Binding Domain (RBD) of the SARS-CoV-2 Spike protein as described (https://doi.org/10.1101/2021.07.09.21260266)..

ELIGIBILITY:
Inclusion Criteria:

* Dental healthcare workers (DHCW)s employed at Rutgers School of Dental Medicine

Exclusion Criteria:

* Previous participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Feldman, DMD, MBA, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
If the COVID test results show that a participant is positive for COVID-19, the study staff will tell the participant the results. The study staff will be required to give the participant's name to the state's Department of Public Health if the participant tests positive because this is the law.
  At the end of the study, de-identified data will be provided to the National Coordinating Center.

REFERENCES:
- [Background] 1. American Dental Association COVID-19 Toolkit - Update to Office Procedures During COVID-19. https://www.ada.org/-/media/project/ada-organization/ada/ada-org/files/resources/coronavirus/update_to_office_procedures_during_covid19.pdf accessed on November 11, 2021.
- [Background] Estrich CG, Mikkelsen M, Morrissey R, Geisinger ML, Ioannidou E, Vujicic M, Araujo MWB. Estimating COVID-19 prevalence and infection control practices among US dentists. J Am Dent Assoc. 2020 Nov;151(11):815-824. doi: 10.1016/j.adaj.2020.09.005. PMID 33071007
- [Background] Shirazi S, Stanford CM, Cooper LF. Testing for COVID-19 in dental offices: Mechanism of action, application, and interpretation of laboratory and point-of-care screening tests. J Am Dent Assoc. 2021 Jul;152(7):514-525.e8. doi: 10.1016/j.adaj.2021.04.019. Epub 2021 May 4. PMID 34176567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 asymptomatic DHCWs in the Oral Medicine clinic, Rutgers School of Dental Medicine, with no history of documented COVID-19 infection or viral exposure, were enrolled. Study participation ranged from January- February 2021.
Groups:
- SARS-CoV-2 Testing: There is only one arm in this study- the study is a non-randomized pilot. All the subjects will be tested for SARS CoV 2 viral Antigen and antibody to the virus as described.
  Testing for SARS CoV2 Antigen and Antibody: Antigen testing: Rapid Antigen testing (Point-of-care) Antibody testing: ELISA testing of microsampling 'finger-prick' specimen DHCW Survey for the adoption of risk mitigation practices and for perceptions of safety
Period: Overall Study
Arm/Group | SARS-CoV-2 Testing
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dental Health Care Worker (DHCW) Willingness to Participate in the Study
Description: Number of Dental Health Care Workers (DHCWs) approached to enroll 10 consenting subjects to participate in the study
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: DHCW Willingness/Ability to Follow Through With the Study Surveys, Triage and Testing
Description: Percentage of Dental Healthcare workers (DHCW)s who complete the study steps of surveys, triage and testing
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 10

3. Primary Outcome: DHCW Test Completion
Description: Percentage of DHCWs with completed SARS-CoV-2 test completed
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 10

4. Primary Outcome: DHCW Ease of Complying With Protocol
Description: Number of DHCWs who reported ease of complying with protocol as their choices on questions on the survey enquiring ease at start-of-study, end-of-study
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 9

5. Primary Outcome: Number of DHCW With Complete Surveys
Description: Number of participants with complete Start-of-study, Triage and End-of-Study surveys
Time Frame: Through study completion (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 10

6. Secondary Outcome: SARS CoV2 Rapid Antigen Testing (Point-of-care)- Number of Participants Who Tested Positive
Description: Number of participants testing positive for SARS CoV2 using a point-of-care Rapid Antigen Testing
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 0

7. Secondary Outcome: Positive Antibody Testing
Description: Number of participants who tested positive for antibody to SARS-CoV2
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 5

8. Secondary Outcome: Number of DCHWs Who Reported Feeling Safe and Comfortable Reporting to Work
Description: Percentage of dental healthcare workers who responded feeling safe and comfortable reporting to work in the survey presented in the pilot study
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 1 month
Description: This study only involved a nasal swab, a finger-prick and survey.
Arm/Group | SARS-CoV-2 Testing
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT05607147/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT05607147/ICF_001.pdf